CLINICAL TRIAL: NCT01156155
Title: Periodontal Disease and P. Gingivalis in Rheumatoid Arthritis
Status: Completed | Type: Observational
Sponsor: University of Nebraska (Other)
Collaborators: Dallas VA Medical Center (U.S. Federal Agency); Washington D.C. Veterans Affairs Medical Center (U.S. Federal Agency); VA Salt Lake City Health Care System (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: 0342-10-FB
Record Dates: First submitted 2010-06-30; First posted 2010-07-02 (Estimated); Last update posted 2023-11-02 (Actual); Status verified 2023-10

CONDITIONS: Rheumatoid Arthritis; Osteoarthritis; Periodontal Disease
Keywords: rheumatoid arthritis; osteoarthritis; periodontal disease
MeSH Terms: conditions — Arthritis, Rheumatoid; Osteoarthritis; Periodontal Diseases | interventions — Blood Specimen Collection; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood specimens (serum, plasma and DNA)will be collected during a one time visit. Also bacterial samples will be collected from the gums of the subject's mouth.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Participants with Rheumatoid Arthritis: Rheumatoid arthritis patients Digital xray of jaw and teeth Blood draw questionnaires Periodontal Examination Bilateral digital xray of hands
  Interventions: Radiation: Digital xray of jaw and teeth; Procedure: Blood draw; Other: questionnaires; Procedure: Periodontal Examination; Other: Bilateral digital xray of hands
- Osteoarthritis: Osteoarthritis patients Digital xray of jaw and teeth Blood draw questionnaires Periodontal Examination
  Interventions: Radiation: Digital xray of jaw and teeth; Procedure: Blood draw; Other: questionnaires; Procedure: Periodontal Examination

INTERVENTIONS:
Radiation: Digital xray of jaw and teeth — one time xray of jaw and teeth
Procedure: Blood draw — Three to four tablespoons of blood drawn.
Other: questionnaires — completed questionnaires regarding patient's health and functional ability.
Procedure: Periodontal Examination — Periodontal examination including measurement of gum pockets with a probe. Bacterial samples taken.
Other: Bilateral digital xray of hands — One time digital xray of hands
  Groups: Participants with Rheumatoid Arthritis

SUMMARY:
Periodontitis (PD) has been postulated to be a risk factor for the onset and progression of rheumatoid arthritis (RA). Recent reports suggest that infection with Porphyromonas gingivalis (P. gingivalis), a major oral pathogen in PD, could play a pivotal role in the development RA. The objective of this study is to examine the relationship of PD and P. gingivalis infection with the risk and severity of RA.

DETAILED DESCRIPTION:
In this study, we will examine whether periodontitis (PD) and P. gingivalis impact rheumatoid arthritis (RA) risk by enrolling 300 patients with RA and 300 comparator patients with osteoarthritis and comparing results from comprehensive dental examinations and antibody responses to P. gingivalis. We will examine whether these associations are modified by the presence of certain genetic risk factors previously implicated in RA and whether evidence of infection with P. gingivalis precedes RA onset by examining banked sera from the Department of Defense Serum Repository (DoDSR) and the Studies of the Etiology of RA (SERA). We also plan to explore whether there are novel proteins expressed by P. gingivalis that drive autoimmunity in RA and whether immune responses to these bacterial proteins predict the future development of RA.

ELIGIBILITY:
Inclusion Criteria:

* Age 19 years or older
* Diagnosis of rheumatoid arthritis, or osteoarthritis
* Have 9 or more evaluable posterior teeth (out of a total of 28 teeth, excluding third molars)
* Willing and able to provide informed consent

Exclusion Criteria:

* Received tetracyclines within the last 6 months.
* Need for antibiotic premedication for dental probing.
* Pregnant or breast feeding

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: UNebraskapatients Omaha VA Medical Center
Sampling Method: Non-Probability Sample
Enrollment: 617 (Actual)
Dates: Start 2010-07-14 (Actual); Primary Completion 2018-08-30 (Actual); Study Completion 2018-08-30 (Actual)

PRIMARY OUTCOMES:
Show the associations of periodontitis with RA are primarily due to infection with P. gingivalis | within thirty days of enrollment
  Clinically defined PD will be more common in RA patients than in controls. 1.B.: Clinically defined PD will be associated with greater RA disease severity including autoantibody status and the presence and extent of radiographic disease progression.
  1.C.: The associations of clinically defined PD with RA risk and severity will be explained by the presence of antibody to P. gingivalis.

CONTACTS AND LOCATIONS:
Overall Officials: Ted R Mikuls, MD, MSPH, Principal Investigator — University of Nebraska
Locations (1):
- Veterans Affairs Medical Center, Omaha, Omaha, Nebraska, United States